CLINICAL TRIAL: NCT05019807
Title: To Compare the Compliance, Knowledge/Awareness About Diabetes, Physical Activity, Diet Plan and Attendance in Patients With Diabetic Macular Edema
Brief Title: Comparing the Compliance to Follow-up in Patients With Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lions Club International Foundation (Other)
Responsible Party: Principal Investigator, Rajiv Raman, Ophthalmologist, Lions Club International Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 864-2020-P
Record Dates: First submitted 2021-08-06; First posted 2021-08-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp group (Other): The arm receives education information about diabetes and its complications, diet and physical activities through WhatsApp.
  Interventions: Other: WhatsApp group
- Control group (Other): The arm does not received any education information.
  Interventions: Other: Control group

INTERVENTIONS:
Other: WhatsApp group — Patients under intervention group will attend an education sessions by structured videos and images with the help of digital tool-WhatsApp group chat administered by the researcher. The group will have the objective interaction with patients and researchers to convey about their view of opinion on sight threatening diabetic retinopathy and management. The structured programme included definition of diabetes mellitus, symptoms, risk factors, awareness of DM and DR, importance of self-care about the disease (eye care and blood glucose monitoring), dietary management and importance of physical activity (Life style modification). The groups will be tracked frequently by WhatsApp/telephonic call and will be documented. Confidentiality of all participants will be maintained.
  Arms: WhatsApp group
Other: Control group — Patient under non-intervention group will not attend or take part in the education sessions or interaction with other patients. Will receive only the general instructions or advises from ophthalmologists about management and follow-up visit.
  Arms: Control group

SUMMARY:
Diabetic retinopathy (DR) is the microvascular complication in the eye due to uncontrolled diabetes. According to the International Diabetes Federation (IDF), 382 million people had diabetes in 2013 and this number is expected to rise to 592 million by 2035, while 175 million people remain undiagnosed. Ninety percent of these people suffer from type 2 Diabetes mellitus(DM). Over time, patients with non-proliferative DR may progress to more advance stages of DR, with increased risk of vision threatening conditions such as diabetic macular edema (DME). DME is the most frequent cause of vision loss in patients with diabetes and eventually can lead to blindness. The management strategy is crucial to prevent or limit the progression of DR. Patient education creates an important tool to control diabetes, to prevent complications and to reduce the cost. Several studies point out that diabetes group education, compared with individual education, was equally effective at improving diabetes control. Another group based education for type 2 DM shown effective in improving HbA1c, knowledge of diabetes, reduction of systolic blood pressure, body weight and requirement for diabetes medication. Studies have showed that group education had significant changes compared with individual education in HbA1c in 6 and 12, months and significant changes were found in fasting blood glucose in 12 months, diabetes knowledge, and self-management skills. Moreover, a study supported that, compared with individual counselling, group self-management education was associated with fewer acute complications and some improvements in the care process. There is no adequate evidence of which educations methods are the most effective in improving clinical outcomes of people with type 2 diabetes. There was a lack in diabetes management in India regarding the multidisciplinary diabetic intervention tool.

Thus the investigator's aim is to focus on interventions to improve the compliance, knowledge/awareness about diabetes, physical activity, diet plan and attendance for diabetic check-up which got emerged from a qualitative study. There is a need to monitor the diabetic patients closely to ensure the compliance towards intervention given at home.

DETAILED DESCRIPTION:
This is a single centre hospital based randomized interventional study. Patients meeting the inclusion criteria will be recruited by researcher, from retina clinic through ophthalmologist who are specialized in diabetic eye examination. The study participants chosen randomly will be given awareness or education by digital tool through smart phone in the intervention group and other half will receive the normal care (non-intervention group). All patients will take their prescribed diabetes medicines as per advised by the diabetologist/physician.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 50 years
* Diagnosed care of DME who had not underwent treatment elsewhere
* Received at least one laser treatment or pharmacotherapy
* Attended at least one follow-up clinical visit
* Patients willing to learn, listed to others and talk about themselves.
* Patients who have access to smart phone.

Exclusion Criteria:

* Patients with ocular co-morbidities other than DME
* Patients refusing to abide by group guidelines and demonstrating serious problems with interpersonal relationships.
* Contrary to popular opinion, people who do poorly in groups.
* Difficult patients who are self-centered.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Follow-up rate in patients with diabetic macular edema receiving education materials about diabetes and its complications. | 12 months
  To investigate the compliance of diabetes management in patients diagnosed with diabetic macular edema after providing educational materials in WhatsApp and compare with control group in a tertiary eye care institute in South India.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Raman, MS,DNB, FRCS"Ed, Principal Investigator — Sankara Nethralaya
Locations (1):
- Rajiv Raman, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the study are not publicly available, as it against the organization hospital policy. But are available from the corresponding author on reasonable request.